CLINICAL TRIAL: NCT04024488
Title: IMPAACT 2016 - Evaluating a Group-Based Intervention to Improve Mental Health and Antiretroviral Therapy (ART) Adherence Among Youth Living With HIV in Low Resource Settings
Brief Title: Group-Based Intervention to Improve Mental Health and Adherence Among Youth Living With HIV in Low Resource Settings
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMPAACT 2016; DAIDS ID #38506 (Other: DAIDS/NIAID/NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: HIV-1-infection
Keywords: Mental Health; Adherence; Trauma-Informed Cognitive Behavioral Therapy
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In the Randomized Trial, youth participants will be randomized in a 1:1 ratio with their caregivers to one of two study arms. One arm is the TI-CBT intervention arm: six 2-hour TI-CBT group sessions lead by Indigenous Youth Leaders (IYL) during weeks 1 - 6 and one 2-hour booster group session at 6-months. The caregivers participating for youth who are enrolled into the TI-CBT arm will receive two 2-hour group sessions led by adult study staff during weeks 1-6 and one 2-hour booster group session at 6-months.
  The other arm is the discussion control arm consisting of: six 2 hour discussion group sessions lead by IYL during weeks 1-6 and one 2-hour booster discussion group session at 6 months. The caregivers of youth randomized to the discussion control arm will have two 2-hour discussion group sessions led by adult study staff during weeks 1-6 and one 2-hour booster discussion group session at 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TI-CBT Intervention Arm (Experimental): In the Randomized Trial, youth participants will be randomized in a 1:1 ratio with their caregivers to one of two study arms. One arm is the TI-CBT intervention arm consisting of: six 2-hour TI-CBT group sessions lead by Indigenous Youth Leaders (IYL) during weeks 1 - 6 and one 2-hour booster group session at 6-months. The caregivers (willing to participate with youth permission) for youth who are enrolled into the TI-CBT arm will be enrolled onto the same arm, and receive two 2-hour group sessions led by adult study staff during weeks 1-6 and one 2-hour booster group session at 6-months. The youth and caregiver sessions are held separately.
  Interventions: Behavioral: TI-CBT Intervention Arm
- Discussion Control Arm (Active Comparator): Arm two is the discussion control arm consisting of: six 2 hour discussion group sessions lead by IYL during weeks 1-6 and one 2-hour booster discussion group session at 6 months. The caregivers (willing to participate with youth permission) for youth randomized to the discussion control arm will have two 2-hour discussion group sessions led by adult study staff during weeks 1-6 and one 2-hour booster discussion group session at 6 months. The youth and caregiver sessions are held separately.
  Interventions: Behavioral: Discussion Control Arm

INTERVENTIONS:
Behavioral: TI-CBT Intervention Arm — TI-CBT teaches techniques and ways to manage distress through psychosocial health education, cognitive restructuring, and "mastery of trauma", which refers to the process by which survivors of psychological trauma work through the traumatic experience in a meaningful way, and are able to move on with life. TI-CBT addresses both the trauma of learning one has HIV and the trauma associated with managing a chronic and stigmatized illness. The intervention highlights links between HIV and traditional gender roles, gender inequities, and gender based violence. Finally, the relaxation training teaches youth strategies to relax and these are integrated at the beginning and end of each session. TI-CBT Youth and Caregiver Intervention Manuals are distributed to sites for translation, backtranslation, and cultural adaptation in preparation for the Randomized Trial.
  Arms: TI-CBT Intervention Arm
Behavioral: Discussion Control Arm — Each youth discussion control group session will be led by IYL and each caregiver discussion control group will be led by adult study staff. Discussion topics will be selected by youth and caregivers in the group as applicable. Discussion Control group session will take place at a separate time from TI-CBT youth group sessions in attempt to minimize contamination. To note, participant and caregiver group sessions are always held separately.
  Arms: Discussion Control Arm

SUMMARY:
IMPAACT 2016 is a multi-site, two-arm, individually randomized, controlled study to evaluate whether an Indigenous Leader Outreach Model (ILOM) of trauma-informed cognitive behavioral therapy (TI-CBT) delivered by Indigenous Youth Leaders (IYL) is associated with improved mental health outcomes and ART adherence among youth living with HIV in resource-limited settings. The intervention is adapted to the local context through advance conduct of focus groups and pilot testing.

DETAILED DESCRIPTION:
IMPAACT 2016 is a multi-site, two-arm, individually randomized, controlled study to evaluate whether an Indigenous Leader Outreach Model (ILOM) of trauma-informed cognitive behavioral therapy (TI-CBT) delivered by Indigenous Youth Leaders (IYL) is associated with improved mental health outcomes and ART adherence among youth living with HIV in resource-limited settings. To adapt the intervention for the local context, the trial will be preceded by an adaption of the TI-CBT intervention at each site using the "ADAPT-ITT" model, which includes focus groups and pilot tests. In the randomized study, youth will be individually randomized to either the TI-CBT Intervention Arm or the Discussion Control Arm. Participants will meet as a group within their randomized arm and receive multiple group sessions within an eight-week period. Each group will include an average of eight youth for an approximate total of 192-256 youth in the Randomized Trial (96-128 youth per arm). TI-CBT and Discussion Control groups in each arm will be mixed-gender unless it is determined necessary to have single-gender groups during the focus group. Caregivers (as available and with youth permission) will be assigned to the same study arm as their youth. Caregivers will meet as a group for two caregiver-specific sessions on two separate weeks and separate from their youth group sessions. Youth and caregivers will complete a follow-up visit immediately after their last group session and two additional follow-up visits at six and 12 months. Youth and caregivers will also receive one two-hour booster group session consistent with their assigned study arm immediately after the six-month evaluations. The booster sessions are intended to enhance treatment effects and increase sustainability. Once all participants have completed their six-month evaluations, data from these evaluations will be analyzed to determine the short-term effects of the intervention. Additional analyses to assess the longer-term effects of the intervention, including the effects of the booster group session, will be performed after the completion of follow-up.

ELIGIBILITY:
Inclusion Criteria - For Youth Participants:

* At screening, 15-19 years old.
* If of legal age to provide independent informed consent as determined by site Standard Operating Procedures (SOPs) and consistent with site IRB/EC policies and procedures: potential youth participant is willing and able to provide written informed consent for study participation.
* If not of legal age to provide independent informed consent: Parent or guardian is willing and able to provide written informed consent for study participation and potential youth participant is willing and able to provide written informed assent for study participation.
* Confirmed HIV-infection based on documented testing of two samples collected at different time points as documented in medical records or by confirmatory testing.
* At screening, aware of his or her HIV infection, as confirmed by Investigator of Record or designee.
* At screening, has been prescribed ART for a minimum of 24 weeks prior to screening based on medical record documentation.
* At screening, meets at least one of the following indicators of moderate to severe mental health symptomology:

  * Patient Health Questionnaire-9 (PHQ-9) score ≥ 10
  * General Anxiety Disorder-7 (GAD-7) score ≥ 10
  * UCLA Post-Traumatic Stress Disorder-Reaction Index (UCLA PTSD-RI) score > 35

Inclusion Criteria - For Caregiver Participants:

* Caregiver, defined as a biological parent, legal guardian, or person who provides emotional, psychological and/or informational care to a youth taking part in the Randomized Trial, as identified by the youth, and for whom the youth has provided written permission to participate in the study.
* Of legal age to provide independent consent and willing and able to provide written informed consent for study participation.

Exclusion Criteria - For Youth Participants:

* At entry, participating in a study delivering a mental health or ART adherence intervention.
* Has prior participation in an IMPAACT 2016 Focus Group or Pilot Test
* Any other condition, adverse social situation or cognitive impairment that, in the opinion of the site investigator, would preclude informed assent and informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Exclusion Criteria - For Caregiver Participants:

Has prior participation in an IMPAACT 2016 Focus Group or Pilot Test.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | at 6-months
  (PHQ-9, measure of depression: range 0-27, higher=worse)
General Anxiety Disorder-7 | at 6-months
  (GAD-7, measure of anxiety: range 0-21, higher=worse)
UCLA Post-Traumatic Stress Disorder-Reaction Index | at 6-months
  (UCLA PTSD-RI, measure of TPSD: range 0-51, higher=worse)
Composite mental health measure | at 6-months
  (measure of combined mental health issues: PHQ-9, GAD-7, and UCLA PTSD-RI scores will be standardized to have mean=0, standard deviation=1, and then summed; higher=worse)

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | after initial treatment completion (an average of 6 weeks)
  (PHQ-9, measure of depression: range 0-27, higher=worse)
General Anxiety Disorder-7 | after initial treatment completion (an average of 6 weeks)
  (PHQ-9, measure of depression: range 0-27, higher=worse)
UCLA Post-Traumatic Stress Disorder-Reaction Index | after initial treatment completion (an average of 6 weeks)
  (UCLA PTSD-RI, measure of TPSD: range 0-51, higher=worse)
Composite mental health measure | after initial treatment completion (an average of 6 weeks)
  (measure of combined mental health issues: PHQ-9, GAD-7, and UCLA PTSD-RI scores will be standardized to have mean=0, standard deviation=1, and then summed; higher=worse)
ART Adherence | after initial treatment completion (an average of 6 weeks), and at 6-months
  Self-report - Wilson 3-item scale (range 0-100, higher=better)
Viral Load | after initial treatment completion (an average of 6 weeks), and at 6-months
  HIV-1 RNA

CONTACTS AND LOCATIONS:
Overall Officials: Geri Donenberg, PhD, Study Chair — University of Illinois at Chicago; Dorothy Dow, MD, MSc, Study Chair — Duke University; Suad Kapetanovic, MD, Principal Investigator — University of Southern California
Locations (8):
- Botswana (2):
  - Gaborone Prevention/Treatment Trials CRS 12701, Gaborone
  - Molepolole Prevention/Treatment Trials CRS 12702, Molepolole
- Malawi (2):
  - College of Medicine CRS 30301, Blantyre
  - University of North Carolina Lilongwe CRS 12001, Lilongwe
- Soweto IMPAACT CRS 8052, Soweto, South Africa
- Zimbabwe (3):
  - St. Mary's CRS 30303, Chitungwiza
  - Harare Family Care CRS 31890, Harare
  - Seke North CRS 30306, Harare

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning three months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  Types of Analyses: Specifically for the types of analyses needed to achieve aims in the proposal approved by the IMPAACT Network.
  Mechanism: Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- See also: IMPAACT 2016 web page — https://www.impaactnetwork.org/studies/impaact2016